CLINICAL TRIAL: NCT02623374
Title: Menopause at Work: Improving the Experience of Menopause for Working Women
Brief Title: MENOS@Work Trial: A Self-help CBT Intervention for Working Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of Nottingham (Other); Wellbeing of Women (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WOW-RG1701
Record Dates: First submitted 2015-11-25; First posted 2015-12-07 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2015-12

CONDITIONS: Menopause

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SH-CBT (Experimental): This intervention will be a tailored CBT intervention adapted from the previously validated (Ayres, et al., 2012) self-help CBT intervention that comprises of a self-help booklet containing information, advice, a relaxation CD and daily diaries. This intervention lasts 4 weeks (approx. 4 hours per week) and the materials guide the individual through each chapter and exercise, including the homework set out for each chapter.
  Interventions: Behavioral: self-help CBT intervention (SHCBT)
- No Treatment-Wait Control (NTWC) (No Intervention): Women will be offered no intervention but will complete questionnaires at the same assessment points as the intervention/treatment arm participant group (i.e. baseline (A0), 6 weeks (A1), 20 weeks (A2) post randomisation). They will be offered the SHCBT intervention off trial following the final assessment (i.e. A2).

INTERVENTIONS:
Behavioral: self-help CBT intervention (SHCBT) — See 'Arms' section
  Arms: SH-CBT

SUMMARY:
The study will be a randomised controlled trial (RCT) of a brief self-help CBT intervention (SHCBT), compared with a no treatment-wait control (NTWC) who do not receive the intervention, on the impact of hot flushes experienced by menopausal women in work settings. The study involves samples from a minimum of two large employers (who have already expressed an interest in taking part) and randomly allocating at least 50 eligible women to the SHCBT intervention and another 50 to a NTWC condition (i.e. a minimum of 100 participants in total). Both groups will complete baseline questionnaires (A0), and follow up assessments at 6 weeks (A1) and 20 weeks (A2) post-randomisation. Questionnaires will be completed online or paper and pencil, providing data on the outcomes of interest to assess the interventions effectiveness and feasibility. Participants of the treatment group will also be invited to take part in an evaluation interview at A2. The NTWC will be offered the intervention off-trial.

DETAILED DESCRIPTION:
While some women go through the menopause without any problems, about 25% have troublesome symptoms that affect their daily lives. Hot flushes and night sweats are the main menopausal symptoms and cause physical discomfort, embarrassment and interfere with sleep. Menopausal symptoms have also been reported as problematic by women when at work. In the UK there are over 3.5 million working women aged between 50 and 65 (the majority of whom will be in the menopause transition or postmenopause), yet there is a general lack of awareness about menopause in work settings. Some women take hormone replacement therapy (HRT) to help them to manage working life, but many prefer non-medical options. While there are effective non-medical interventions (such as cognitive behaviour therapy) to help women to manage and cope with menopausal symptoms, these are not yet widely available on the NHS or in the workplace.

In a recent study of 896 women's experiences of working through the menopausal transition in the UK, Griffiths and colleagues (2013) found that the menopausal transition caused difficulties for them, mainly due to troublesome hot flushes, poor concentration, tiredness, poor memory, feeling low/depressed and lowered confidence. Some women were also concerned that their work performance had been negatively affected. Those who were taking HRT did so mainly to help them to cope at work but over 30% of these had side effects or felt that HRT had not helped. The majority of women were unwilling to disclose menopause-related health problems to line managers, most of whom were men or younger than them. Four major areas of need were identified: (i) greater awareness among managers about menopause as a possible occupational health issue, (ii) flexible working hours, (iii) access to information and sources of support at work, and (iv) attention to workplace temperature and ventilation. The authors concluded that employers should be aware that menopausal transition can cause difficulty for some women at work, and that much can be done to support them. The proposed research will aim to target (iii).

Hunter and colleagues (2012) have developed a brief non-medical treatment to help women to manage hot flushes and night sweats, based on cognitive behaviour therapy (CBT), to help women to manage menopausal symptoms. They have evaluated group and self-help forms of the interventions, and found them to be highly effective in reducing how problematic the symptoms are rated. Women receive information and advice to help them to develop strategies to reduce stress, to deal with hot flushes and to improve sleep disrupted by night sweats. In recent randomised controlled trials, women who received the CBT intervention benefited from improvements in hot flushes and night sweats, sleep and perception of memory and concentration, and ability to cope, resulting in benefits to quality of life compared to those who received usual care. Interestingly, the self-help CBT (containing the same information in a booklet with a relaxation CD) was as effective as the group CBT.

The proposed research builds upon these findings and aims to develop and examine the feasibility and impact of an adapted self-help CBT intervention (SHCBT) based on Hunter's early work to help management symptoms and improve the quality of life for working menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Employed women aged 45-60 years
* Have at least 10 problematic (score >2 on HFRS) hot flushes per week for at least two months
* Have a good understanding of English

Exclusion Criteria:

* Men
* Women who cannot understand English
* Women with problematic mental health conditions that may affect participation in the study
* Women not employed (by participating organisations)
* Women outside the inclusion age range and symptom criteria.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Problematic hot flushes | Measurements will be taken at A1 (6 weeks postrandomisation).
  Measured using the Hot Flush Rating Scale (HFRS) by Hunter & Liao (1995), which includes a score between 1-10 based on the mean of three 3-point Likert scales (1=no problem at all, 10=very much a problem) assessing hot flushes and night sweats (HFNS) bother, interference, and distress.
Problematic hot flushes | Measurements will be taken at A2 (20 weeks postrandomisation).
  Measured using the Hot Flush Rating Scale (HFRS) by Hunter & Liao (1995), which includes a score between 1-10 based on the mean of three 3-point Likert scales (1=no problem at all, 10=very much a problem) assessing hot flushes and night sweats (HFNS) bother, interference, and distress.

SECONDARY OUTCOMES:
Problematic hot flushes (frequency) | Measurements will be taken at A1 (6 weeks postrandomisation).
  Measured using the Hot Flush Rating Scale (HFRS) by Hunter & Liao (1995), which gives provides a retrospective recording of the frequency of HFNS and the average severity of the HFNW for the previous week (1=mild, 2=moderate, 3=severe).
Problematic hot flushes (frequency) | Measurements will be taken at A2 (20 weeks postrandomisation).
  Measured using the Hot Flush Rating Scale (HFRS) by Hunter & Liao (1995), which gives provides a retrospective recording of the frequency of HFNS and the average severity of the HFNW for the previous week (1=mild, 2=moderate, 3=severe).
Menopause Representation Questionnaire (Hunter & O'Dea, 2001) | Measurements will be taken at A1 (6 weeks postrandomisation).
  designed to assess women's attributions (identity) of symptoms to the menopause (20 items) and beliefs subscales (cognitive representations) about the menopause (17 items). The belief items are scored on 5-point scales from strongly agree (5) to strongly disagree (1), and mean scores are calculated for beliefs subscales. The identity subscale items are scored from 0 to 2 and summed.
Menopause Representation Questionnaire (Hunter & O'Dea, 2001) | Measurements will be taken at A2 (20 weeks postrandomisation).
  designed to assess women's attributions (identity) of symptoms to the menopause (20 items) and beliefs subscales (cognitive representations) about the menopause (17 items). The belief items are scored on 5-point scales from strongly agree (5) to strongly disagree (1), and mean scores are calculated for beliefs subscales. The identity subscale items are scored from 0 to 2 and summed.
Attitude to Menopause at Work | Measurements will be taken at A1 (6 weeks postrandomisation).
  This measures attitude to menopause and work and whether women feel that their job performance has been affected by menopausal symptoms, and whether they feel that menopause has negatively affected manager's and colleagues views of competence at work (Griffiths, et al., 2010). Contains 2 items scored on 5-point scales (agree (5) to strongly disagree (1)).
Attitude to Menopause at Work | Measurements will be taken at A2 (20 weeks postrandomisation).
  This measures attitude to menopause and work .e. whether women feel that their job performance has been affected by menopausal symptoms, and whether they feel that menopause has negatively affected manager's and colleagues views of competence at work (Griffiths, et al., 2010). Contains 2 items scored on 5-point scales (agree (5) to strongly disagree (1)).
Hot Flush and Night Sweats Belief & Behaviour | Measurements will be taken at A1 (6 weeks postrandomisation).
  16 items to measure beliefs about hot flushes and night sweats (HFNS) and behavioural reactions to cope with HFNS using a 6-point scale from strongly disagree (0) to strongly agree (5). This is a shortened and combined version of Hot Flush Belief & Behaviour Scale (Rendall, et al, 2008; Hunter et al, 2011)
Hot Flush and Night Sweats Belief & Behaviour | Measurements will be taken at A2 (20 weeks postrandomisation).
  16 items to measure beliefs about hot flushes and night sweats (HFNS) and behavioural reactions to cope with HFNS using a 6-point scale from strongly disagree (0) to strongly agree (5). This is a shortened and combined version of Hot Flush Belief & Behaviour Scale (Rendall, et al, 2008; Hunter et al, 2011)
Presenteeism (Koopman et al, 2002) | Measurements will be taken at A1 (6 weeks postrandomisation).
  Stanford Presenteeism Scale (SPS6, Koopman, et al 2002) is used to measure workplace presenteeism, comprises of 6 items that are summed to produce a total presenteeism score. Each item asks the respondent to indicate their work experience over the last month using a 5-point scale (1=strongly disagree, 5=strongly agree).
Presenteeism (Koopman et al, 2002) | Measurements will be taken at A2 (20 weeks postrandomisation).
  Stanford Presenteeism Scale (SPS6, Koopman, et al 2002) is used to measure workplace presenteeism, comprises of 6 items that are summed to produce a total presenteeism score. Each item asks the respondent to indicate their work experience over the last month using a 5-point scale (1=strongly disagree, 5=strongly agree).
Workplace absence (duration) | Measurements will be taken at A1 (6 weeks postrandomisation).
  Participants asked to provide detail of number of days they have taken off from work over the last 4 weeks because of the menopause.
Workplace absence (duration) | Measurements will be taken at A2 (20 weeks postrandomisation).
  Participants asked to provide detail of number of days they have taken off from work over the last 4 weeks because of the menopause.
Workplace absence (spells) | Measurements will be taken at A1 (6 weeks postrandomisation).
  Participants asked to provide detail of average length of spells of absence from work over the last 4 weeks because of the menopause.
Workplace absence (spells) | Measurements will be taken at A2 (20 weeks postrandomisation).
  Participants asked to provide detail of average length of spells of absence from work over the last 4 weeks because of the menopause.
Workplace absence (arriving late/leaving early) | Measurements will be taken at A1 (6 weeks postrandomisation).
  Participants asked to provide detail of any time over the last 4 weeks been late to work of left work early because of the menopause.
Workplace absence (arriving late/leaving early) | Measurements will be taken at A2 (20 weeks postrandomisation).
  Participants asked to provide detail of any time over the last 4 weeks been late to work of left work early because of the menopause.
Menopausal symptom disclosure to manager | Measurements will be taken at A1 (6 weeks postrandomisation).
  Menopausal symptom disclosure to managers is measured using a single dichotomous item ('yes' or 'no'; Griffiths, et al, 2010, 2013) and whether participants have told their manager about any reduced working hours (i.e. arriving late, leaving early) due to their menopausal symptoms (if appropriate) 'yes', 'no', 'sometimes').
Menopausal symptom disclosure to manager | Measurements will be taken at A2 (20 weeks postrandomisation).
  Menopausal symptom disclosure to managers is measured using a single dichotomous item ('yes' or 'no'; Griffiths, et al, 2010, 2013) and whether participants have told their manager about any reduced working hours (i.e. arriving late, leaving early) due to their menopausal symptoms (if appropriate) 'yes', 'no', 'sometimes').
Turnover intentions | Measurements will be taken at A1 (6 weeks postrandomisation).
  Work turnover intentions are measured with 4 items (Shore and Martin, 1980), to assess how likely the individual is to leave their organisation). Each item contains 5 response options indicating low (1) to high (5) intentions to remain in their organisation that can be averaged to provide an overall score. Two further items are used to measure the degree to which the individual has considered reducing their working hours or leaving the workforce altogether ('yes', 'no', 'sometimes').
Turnover intentions | Measurements will be taken at A2 (20 weeks postrandomisation).
  Work turnover intentions are measured with 4 items (Shore and Martin, 1980), to assess how likely the individual is to leave their organisation). Each item contains 5 response options indicating low (1) to high (5) intentions to remain in their organisation that can be averaged to provide an overall score. Two further items are used to measure the degree to which the individual has considered reducing their working hours or leaving the workforce altogether ('yes', 'no', 'sometimes').
Job satisfaction | Measurements will be taken at A1 (6 weeks postrandomisation).
  A single-item 7-point Likert scale (1=extremely dissatisfied, 4=neither dissatisfied or satisfied, 7=extremely satisfied) to indicate an individual's level of contentment with their job (Griffiths et al, 2010,2013).
Job satisfaction | Measurements will be taken at A2 (20 weeks postrandomisation).
  A single-item 7-point Likert scale (1=extremely dissatisfied, 4=neither dissatisfied or satisfied, 7=extremely satisfied) to indicate an individual's level of contentment with their job (Griffiths et al, 2010,2013).
Job performance | Measurements will be taken A1 (6 weeks postrandomisation).
  A single self-report item. Participants are asked to rate their performance compared to others in a similar role or position to themselves usinf a 5-point Likert scale (1=poor, 5=excellent).
Job performance | Measurements will be taken A2 (20 weeks postrandomisation).
  A single self-report item. Participants are asked to rate their performance compared to others in a similar role or position to themselves usinf a 5-point Likert scale (1=poor, 5=excellent).
Job stress | Measurements will be taken at A1 (6 weeks postrandomisation).
  A single, self-report item asking participants to indicate on a 4-point Likert scale how stressful they find their job (1=not stressful, 4=extremely stressful) (Houdmont et al, 2012).
Job stress | Measurements will be taken at A2 (20 weeks postrandomisation).
  A single, self-report item asking participants to indicate on a 4-point Likert scale how stressful they find their job (1=not stressful, 4=extremely stressful) (Houdmont et al, 2012).
Perceptions of physical and emotional menopausal symptoms | Measurements will be taken at A1 (6 weeks postrandomisation).
  Women's Health Questionnaire (Hunter, 1992) used to assess participant perceptions of symptoms using a 4-point Likert scale. Includes 37 items.
Perceptions of physical and emotional menopausal symptoms | Measurements will be taken at A2 (20 weeks postrandomisation).
  Women's Health Questionnaire (Hunter, 1992) used to assess participant perceptions of symptoms using a 4-point Likert scale. Includes 37 items.
Sleep quality (Mundt, et al, 2002) | Measurements will be taken at A1 (6 weeks postrandomisation).
  Single item from Pittsburgh Sleep Quality Index (PSQI) (Buysse et al., 1989) that measures quality of sleep over the last month using a 5-point likert scale (very good=5 to very bad = 1).
Sleep quality (Mundt, et al, 2002) | Measurements will be taken at A2 (20 weeks postrandomisation).
  Single item from Pittsburgh Sleep Quality Index (PSQI) (Buysse et al., 1989) that measures quality of sleep over the last month using a 5-point likert scale (very good=5 to very bad = 1).
Personal resilience at work | Measurements will be taken at A1 (6 weeks postrandomisation).
  Single item that measures participants' self-perceived level of resilience in the work context (Hardy et al, in prep) used using a 9-point scale (1=low resilience to 9=high resilience).
Personal resilience at work | Measurements will be taken at A2 (20 weeks postrandomisation).
  Single item that measures participants' self-perceived level of resilience in the work context (Hardy et al, in prep) used using a 9-point scale (1=low resilience to 9=high resilience).

OTHER OUTCOMES:
Use of medical resources for menopause (visits) | Measurements will be taken at A2 (20 weeks postrandomisation).
  The use of medical resources for menopause and treatments for HFNS will be monitored, to determine how often visited their GP/hospital doctor/nurse about the menopause since starting the trial.
Use of medical resources for menopause (treatments for HFNS) | Measurements will be taken at A2 (20 weeks postrandomisation).
  The use of medical resources for treatments for HFNS will be monitored, by asking whether they have/are currently taking any treatment (medical or non-medical) for HFNS (dichotomous: yes/no).
Adherence, acceptability and feasibility of intervention: completion | Measurements will be taken at A1 (6 weeks postrandomisation).
  Question about how much of the booklet they read using a 4-point likert scale (not at all - all of it).
Adherence, acceptability and feasibility of intervention: completion | Measurements will be taken at A2 (20 weeks postrandomisation).
  Question about how much of the booklet they read using a 4-point likert scale (not at all - all of it).
Adherence, acceptability and feasibility of intervention: changes in coping | Measurements will be taken at A1 (6 weeks postrandomisation).
  Six items using a 5-point Likert scale (1=not at all to 5 =extremely) asking whether the guide has affected their management of dealing with stress and coping in the past 4 weeks.
Adherence, acceptability and feasibility of intervention: changes in coping | Measurements will be taken at A2 (20 weeks postrandomisation).
  Six items using a 5-point Likert scale (1=not at all to 5 =extremely) asking whether the guide has affected their management of dealing with stress and coping in the past 4 weeks.
Adherence, acceptability and feasibility of intervention: relaxation and breathing | Measurements will be taken at A1 (6 weeks postrandomisation).
  4 items using 5-point scales to evaluate the relaxation and breathing exercises.
Adherence, acceptability and feasibility of intervention: relaxation and breathing | Measurements will be taken at A2 (20 weeks postrandomisation).
  4 items using 5-point scales to evaluate the relaxation and breathing exercises.

CONTACTS AND LOCATIONS:
Overall Officials: Myra S Hunter, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

REFERENCES:
- [Derived] Boxall C, Fenlon D, May C, Nuttall J, Hunter MS. Implementing a nurse-delivered cognitive behavioural therapy intervention to reduce the impact of hot flushes/night sweats in women with breast cancer: a qualitative process evaluation of the MENOS4 trial. BMC Nurs. 2023 Sep 15;22(1):317. doi: 10.1186/s12912-023-01441-3. PMID 37715249
- [Derived] Hardy C, Griffiths A, Norton S, Hunter MS. Self-help cognitive behavior therapy for working women with problematic hot flushes and night sweats (MENOS@Work): a multicenter randomized controlled trial. Menopause. 2018 May;25(5):508-519. doi: 10.1097/GME.0000000000001048. PMID 29315132
- [Derived] Hunter MS, Hardy C, Norton S, Griffiths A. Study protocol of a multicentre randomised controlled trial of self-help cognitive behaviour therapy for working women with menopausal symptoms (MENOS@Work). Maturitas. 2016 Oct;92:186-192. doi: 10.1016/j.maturitas.2016.07.020. Epub 2016 Jul 29. PMID 27621258